CLINICAL TRIAL: NCT07317518
Title: The Effect of Different Kinesio Taping Techniques Applied to Patients With Chronic Low Back Pain on the Thoracolumbar Fascia: A Randomized Controlled Trial
Brief Title: The Effect of Different Kinesio Taping Techniques Applied to Patients With Chronic Low Back Pain on the Thoracolumbar Fascia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Safak Kuzu, Assist. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52066301980.
Record Dates: First submitted 2025-12-15; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: Non-specific chronic low back pain; Kinesio taping; Thoracolumbar fascia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Functional Fascial Taping Group): (Experimental): For this group, "I" and "Y" kinesiology tape will be applied using a fascial correction technique on the thoracolumbar fascia with 10-50% oscillatory (oscillating) tension. The taping direction will be determined based on the direction in which pain is most reduced during movement.
  Interventions: Other: Functional Fascial Taping Group; Other: Traditional treatment
- Group 2 (Muscle Technique Taping Group): (Active Comparator): This group will be applied using "I" strip kinesiology tape muscle taping techniques on the paravertebral muscles. Two of the tapes will be applied completely tension-free (0%), while one will be applied transversely to the sacroiliac region with 25% tension.
  Interventions: Other: Muscle Technique Taping Group; Other: Traditional treatment
- Group 3 (Damascus Taping Group): (Sham Comparator): This group will receive kinesiology tape applied symbolically to the skin over the thoracolumbar region without any therapeutic taping technique, without targeting fascia or muscle correction, and without creating meaningful tension (0% tension). Sham taping will be used to control for the placebo effect, independent of the specific mechanical and neurophysiological effects of taping.
  Interventions: Other: Damascus Banding Group; Other: Traditional treatment

INTERVENTIONS:
Other: Functional Fascial Taping Group — The treatment program for the Functional Fascial Taping Group is as follows: Participants in this group will undergo a targeted fascial correction technique applied to the thoracolumbar fascia. In practice, "I" and "Y" strips cut from 5 cm x 5 m kinesiology tape will be used, and the tapes will be applied to the right and left thoracolumbar fascia with an oscillatory (oscillating) tension in the range of 10-50%. The protocol will be repeated for a total of 2 weeks (4 sessions), twice a week, and the tapes will be replaced at each session. The primary goal is to reduce pain and improve function by directly affecting the biomechanics of the fascial tissue. Patients in the stabilization exercises group will perform cervical stabilization exercises consisting of 3 levels with gradually increasing difficulty. The exercises will be taught to patients level by level by a physical therapist over 6 weeks. Stretching exercises will be performed before each exercise session.
  Arms: Group 1 (Functional Fascial Taping Group):
Other: Muscle Technique Taping Group — In this group, the more traditional approach of muscle taping will be adopted. The application will be performed using three "I"-shaped strips of tape. The first two strips will be placed completely tension-free (0%) on the paravertebral muscles while the patient is leaning forward and performing a slight rotation. The third tape will be applied transversally with 25% tension, parallel to the ground, over the sacroiliac joints. This protocol will also be applied twice a week for two weeks, with the aim of providing muscle support and increasing stabilization.
  Arms: Group 2 (Muscle Technique Taping Group):
Other: Damascus Banding Group — The taping applied in this group will not aim to correct any muscles or fascia, will be performed without applying therapeutic tension (0% tension), and will not produce a standard clinical effect. At the end of the study, all participants will be informed that they can access known effective taping approaches upon request.
  Arms: Group 3 (Damascus Taping Group):
Other: Traditional treatment — Patients in the stabilization exercise group will be given cervical stabilization exercises consisting of 3 levels with gradually increasing difficulty. The exercises will be taught to patients level by level by a physical therapist over 6 weeks. Patients will perform the exercises for a total of 6 weeks. Patients will be asked to perform stretching exercises before each exercise session.

SUMMARY:
This study aims to evaluate the effects of functional thoracolumbar fascia kinesiology taping on fascia thickness, pain, and functional disability in individuals with nonspecific chronic low back pain. The study is planned as a randomized controlled trial and will include a total of 30 individuals aged 18-65 years who have been diagnosed with nonspecific mechanical chronic low back pain. Participants will be randomly assigned to two groups: the Functional Fascial Taping Group will receive kinesiology tape applied to the thoracolumbar fascia using a fascia correction technique, while the Muscle Technique Taping Group will receive traditional muscle taping applied to the paravertebral muscles. Interventions will be performed twice a week for two weeks. Assessments will be performed before and after treatment; pain intensity will be measured using the Visual Analog Scale, pressure pain threshold will be measured using an algometer, functional disability will be measured using the Oswestry Low Back Pain Disability Index, and thoracolumbar fascia thickness will be measured using ultrasonography. The findings are expected to contribute to clinical practice by providing evidence-based data on the effectiveness of different kinesiology taping techniques in chronic low back pain.

DETAILED DESCRIPTION:
Non-specific chronic low back pain is a highly prevalent musculoskeletal condition associated with recurrent symptoms, functional limitations, and substantial psychosocial burden. Current clinical practice frequently relies on passive treatment approaches, including various taping techniques; however, the specific effects of different kinesio taping methods on fascial structures remain insufficiently explored. In particular, objective evidence regarding changes in thoracolumbar fascia morphology following targeted taping interventions is limited.

This randomized controlled study aims to compare the effects of functional fascial kinesio taping and conventional muscle taping on thoracolumbar fascia thickness, pain perception, and functional disability in individuals with non-specific chronic low back pain. Participants diagnosed with non-specific mechanical chronic low back pain will be randomly allocated to one of two intervention groups. One group will receive functional fascial taping applied according to movement-based pain modulation principles, while the comparison group will receive traditional muscle-oriented kinesio taping. Both interventions will be administered over a short-term treatment period without additional therapeutic modalities to isolate the effects of taping.

Outcome assessment will focus on changes in pain intensity, pressure pain sensitivity, functional disability, and thoracolumbar fascial characteristics. Fascial thickness will be evaluated using ultrasonographic imaging to provide an objective measure of tissue-level response. By integrating subjective clinical outcomes with imaging-based assessment, this study seeks to clarify whether taping strategies that target fascial mechanics offer advantages over conventional muscle-focused approaches.

The findings are expected to contribute to evidence-based decision-making in rehabilitation practice by informing clinicians about the potential role of fascia-oriented taping in the management of chronic low back pain, while minimizing redundancy with procedural and technical details documented elsewhere in the study record.

ELIGIBILITY:
Inclusion Criteria:

* Age: Be between 18 and 65 years old.
* Volunteer status: Be willing to participate in the study and sign an informed consent form.
* Diagnosis: Have been diagnosed by a physician with nonspecific mechanical chronic low back pain. This diagnosis is defined as follows:
* A pain episode lasting longer than 6 weeks or
* A history of recurrent low back pain (episodes lasting longer than 24 hours with at least one pain-free period of one month before/after the episode).
* Localization: Pain localized between the lowest rib and the gluteal folds.

Exclusion Criteria:

* Specific Spinal Pathologies: The presence of a specific cause for back pain (e.g., structural abnormalities such as herniation, stenosis, spondylolisthesis).
* History of Major Trauma: A history of serious trauma to the back region.
* Systemic Diseases: Systemic diseases that may affect the outcome, such as rheumatological diseases or diabetes.
* History of Cancer: Any cancer diagnosis or history.
* Osteoporosis: Diagnosis of bone loss.
* Inflammatory or Neurological Diseases: Diagnosis of inflammatory rheumatic diseases such as ankylosing spondylitis or a neurological disease.
* Radicular Pain: Presence of radicular pain radiating to the legs, suggesting nerve root compression.

Skin Conditions:

* Known skin sensitivity or allergy to the patches.
* Active dermatitis or pre-existing skin lesion in the patch application area.
* Recent Treatments: Having undergone a physical therapy and rehabilitation (PTR) program targeting the lumbar region or an intervention such as an injection within the last 3 months prior to the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 6 week
  The Visual Analog Scale (VAS) will be used to measure participants' pain intensity. Participants are asked to indicate their current state by placing a line or dot on a 10-centimeter straight line, where both ends are defined by the parameter to be measured in the individual. Pain intensity in the individual is calculated in this way. For example, the parameters to be evaluated are determined at one end of the drawn 10-centimeter straight line (0 = no pain, 10 = unbearable pain).
The thoracolumbar fascia thickness/ULTRASOUND | 6 week
  The thoracolumbar fascia thickness will be measured using the Versana Primer R2 VS GE (China, 2022) ultrasound with a 4.0-13.0 MHz, 38.4 mm probe and a scanning protocol performed at the L3 level of the lumbar spine. Measurements will be performed by an experienced physician doctor in musculoskeletal ultrasound. Measurements will be performed bilaterally in the standard manner, with the patient lying comfortably in the prone position. Measurements will be performed using ultrasound B-mode and a depth setting of 30 mm. Sufficient gel will be used to avoid probe compression on the skin to ensure accurate measurements. To prevent TLF thickness differences from affecting the results, measurements will be taken at 3 separate points and averaged. As recommended by Pirri et al., the probe will be placed perpendicularly, and short and long axis images will be obtained. Images will be recorded and measurements will be taken (Pirri et al., 2024).

SECONDARY OUTCOMES:
LOW BACK PAIN DISABILITY | 6 week
  The Oswestry Back Pain Disability Questionnaire will be used to obtain information about how much back (or leg) pain affects a person's daily activities. The questionnaire consists of 10 sections. The patient is asked to mark the most appropriate answer for themselves. The score is calculated, and the resulting percentage values are interpreted according to the values given below (Yi, 2008); 0% - 20% - minimal disability 20% - 40% - moderate disability 40% - 60% - severe disability 60% - 80% - disabled 80% - 100% - bedridden
Posture | 6 week
  Spinal posture was assessed using a computer-assisted wireless Spinal Mouse device (Spinal Mouse System, Idiag, Fehraltorf, Switzerland). The device was guided manually along the spinous processes from C7 to S3 while the participant stood in a relaxed upright position. The Spinal Mouse records sagittal spinal curvature and calculates numerical values for thoracic kyphosis, lumbar lordosis, and overall spinal inclination. All postural alignment parameters were automatically transferred to the computer software and expressed as angular values (degrees).
Lateral Bridge Testt | 6 week
  The lateral bridge test will be used to evaluate lateral core muscle endurance. Participants will be instructed to lie on their right side, supporting their body on the forearm and feet, with the body aligned in a straight line. The non-supporting arm will rest along the body. Participants will be asked to maintain this position for as long as possible. The test will be terminated when proper alignment is lost or when the pelvis contacts the examination surface. The duration the position is held will be recorded in seconds (Bliss & Teeple, 2005).
Spinal Mobility: | 6 week
  Spinal mobility was evaluated with the same Spinal Mouse system by assessing trunk flexion posture. Participants were instructed to perform maximal trunk flexion from the standing position, and the device was rolled along the spine during the movement. The Spinal Mouse quantitatively measured segmental and total spinal range of motion by calculating angular changes between adjacent vertebral segments. The system provides cumulative numerical values for spinal flexion mobility in degrees. Spinal mobility measurements were recorded at baseline and at the 6-week follow-up.
Postural Endurance (Postural Competence): | 6 week
  Postural endurance was assessed using the Spinal Mouse device during a standardized static loading task. Participants were asked to hold a weight equivalent to 5% of their body weight with both hands at shoulder level, arms parallel to the floor, for 30 seconds while maintaining an upright posture. Immediately after the task, spinal posture was re-measured using the Spinal Mouse. Changes in spinal alignment angles before and after the endurance task were calculated numerically by the software and used as indicators of postural endurance (competence).
Static Trunk Extension Test (Sorensen Test): | 6 week
  The Sorensen test will be performed to assess endurance of the trunk extensor muscles. Participants will lie in a prone position with the pelvis, hips, and knees supported on the examination table, while the upper body extends beyond the edge of the table. The lower extremities will be stabilized by straps or manual fixation. Participants will be instructed to maintain the upper body in a horizontal position with arms crossed over the chest. The test will end when the participant is unable to maintain the horizontal position or reports fatigue. Endurance time will be recorded in seconds (Baltacı et al., 2006).
Trunk Flexor Endurance Test | 6 week
  Trunk flexor endurance will be assessed using a standardized static trunk flexion test. Participants will sit on the examination table with the trunk flexed to approximately 60 degrees, hips and knees flexed, and feet secured. Arms will be crossed over the chest. Participants will be instructed to maintain this position without support for as long as possible. The test will be terminated when the participant is unable to maintain the target position or reports exhaustion. The duration will be measured in seconds using a stopwatch (Bliss & Teeple, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Şafak KUZU, Study Director — Kirsehir Ahi Evran Universitesi

IPD SHARING:
Plan to Share IPD: No